CLINICAL TRIAL: NCT00041821
Title: Individual Factors in Nasal Irritant Sensitivity
Brief Title: Nasal Irritation Study: Individual Factors in Nasal Irritant Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 10424-CP-001
Record Dates: First submitted 2002-07-18; First posted 2002-07-22 (Estimated); Last update posted 2006-03-23 (Estimated); Status verified 2006-03

CONDITIONS: Rhinitis, Allergic, Nonseasonal
Keywords: rhinitis; irritation; trigeminal
MeSH Terms: conditions — Rhinitis, Allergic, Perennial; Rhinitis

INTERVENTIONS:
Procedure: Nasal irritation thresholds and irritant provocation

SUMMARY:
This study seeks to document differences in nasal irritant sensitivity within the population. The investigators are interested in knowing whether age, gender, and allergy status (nasal allergies) predict nasal irritant sensitivity. This is important in understanding symptom reporting patterns in air pollution situations (particularly in so-called "problem buildings"), as well as in understanding the reflex mechanism of a response of the nose to irritants (e.g., nasal congestion).

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* 18-69 years of age
* With or without allergic rhinitis (hay fever)
* In good general health and with no prior history of asthma

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- Upper Airway Biology Laboratory, Richmond, California, United States

REFERENCES:
- [Background] Shusterman DJ, Murphy MA, Balmes JR. Subjects with seasonal allergic rhinitis and nonrhinitic subjects react differentially to nasal provocation with chlorine gas. J Allergy Clin Immunol. 1998 Jun;101(6 Pt 1):732-40. doi: 10.1016/S0091-6749(98)70302-1. PMID 9648699
- [Background] Shusterman D, Murphy MA, Balmes J. The influence of sex, allergic rhinitis, and test system on nasal sensitivity to airborne irritants: a pilot study. Environ Health Perspect. 2001 Jan;109(1):15-9. doi: 10.1289/ehp.0110915. PMID 11171519
- See also: Website of UCSF Upper Airway Biology Laboratory — http://www.noselab.net